CLINICAL TRIAL: NCT05687812
Title: Effects of Cephalaria Syriaca Flour-added Bread on Glucose Metabolism and Appetite Parameters in Individuals With Obesity, Diabetes, and Healthy Controls.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Fulya Calikoglu, MD, PhD; Academician; Principle Investigator, Istanbul University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/342
Record Dates: First submitted 2023-01-08; First posted 2023-01-18 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Nutrition, Healthy
Keywords: Cephalaria Syriaca, glycemic index, type 2 diabetes, obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diabetic group (Experimental): After 10-12 h fasting, an OGTT test with 75 g glucose was performed on the participants, showing no glucose metabolism disorder. Another independent day was chosen as the test day, and the participants were asked to no-restrict carbohydrates and not make any changes in their diet in the days before the test. Volunteers were fed 100g of white bread containing only 250 ml of water and 50g of carbohydrate (CH) for breakfast (after 12 hours of fasting). After 1 week, the same participants were fed 250 ml of water and 100g of test bread (consisting of 0.2% Cephalaria Syriaca flour bread) containing 50g of carbohydrates (KH). During the test, venous and capillary blood samples were taken at 0, 30, 60, 90, and 120 minutes.
  Interventions: Dietary Supplement: Cephalaria Syriaca flour-added bread
- Non-diabetic obese group (Experimental): After 10-12 h fasting, an OGTT test with 75 g glucose was performed on the participants, showing no glucose metabolism disorder. Another independent day was chosen as the test day, and the participants were asked to no-restrict carbohydrates and not make any changes in their diet in the days before the test. Volunteers were fed 100g of white bread containing only 250 ml of water and 50g of carbohydrate (CH) for breakfast (after 12 hours of fasting). After 1 week, the same participants were fed 250 ml of water and 100g of test bread (consisting of 0.2% Cephalaria Syriaca flour bread) containing 50g of carbohydrates (KH). During the test, venous and capillary blood samples were taken at 0, 30, 60, 90, and 120 minutes.
  Interventions: Dietary Supplement: Cephalaria Syriaca flour-added bread
- Non-diabetic and non-obese healthy group (Experimental): After 10-12 h fasting, an OGTT test with 75 g glucose was performed on the participants, showing no glucose metabolism disorder. Another independent day was chosen as the test day, and the participants were asked to no-restrict carbohydrates and not make any changes in their diet in the days before the test. Volunteers were fed 100g of white bread containing only 250 ml of water and 50g of carbohydrate (CH) for breakfast (after 12 hours of fasting). After 1 week, the same participants were fed 250 ml of water and 100g of test bread (consisting of 0.2% Cephalaria Syriaca flour bread) containing 50g of carbohydrates (KH). During the test, venous and capillary blood samples were taken at 0, 30, 60, 90, and 120 minutes.
  Interventions: Dietary Supplement: Cephalaria Syriaca flour-added bread

INTERVENTIONS:
Dietary Supplement: Cephalaria Syriaca flour-added bread — 100g of test bread (consisting of 0.2% Cephalaria Syriaca flour bread) containing 50g of carbohydrates (KH).

SUMMARY:
Cephalaria Syriaca is a common weed in Anatolia and grows wild in wheat fields, with high fat, protein, and dietary fiber content. This study it is aimed to evaluate the effects of lowering the glycemic index of white bread consumed in large quantities in Turkey by adding Cephalaria Syriaca, on healthy, obese, and diabetic individuals.

DETAILED DESCRIPTION:
Nutrition is essential in the treatment and management of diabetes and obesity, and other accompanying diseases. Consumption of low glycemic index (GI) foods is the primary approach in medical nutrition therapy to ensure glycemic control and long-term satiety. The glycemic index is the rate at which foods raise blood sugar. The GI is determined by comparing the area of increase in blood glucose within 2 hours after consumption and absorption of a test food containing 100 g of digestible carbohydrates to the area of increase in glucose generated by the reference food containing the same amount of carbohydrates (primarily white bread). The GI value of the food taken as a reference is 100, and the reference ranges of foods are ≤55 low, 56-69 moderate, and ≥70 high GI. Annual bread consumption is much higher than the world average in Turkey and is about 400 g/day. It has been determined that 66% of the energy consumed per capita is provided from cereals, 56% of this energy is met from bread, and 50% of the protein in the daily diet is completed from bread.

It has been reported that the GI of white bread is 87 in our country and 70 in other countries. Reducing the GI value of a large amount of food consumed will be a positive step for obesity and diabetes management.

Cephalaria syriaca, common in Anatolia and growing wild in wheat fields, has high oil (~20%), protein (15.5%), dietary fiber (25.5%), and polyphenol content and is an annual weed rich in vitamins and minerals. It is known that the flour obtained from Cephalaria Syricia seed strengthens even the flours with low core quality. For this reason, it is used especially in rural areas to increase dough and bread quality. It is known that dietary fiber, fat, and protein contents in foods lower the GI value. Therefore, Cephalaria Syricia flour added to bread flour is expected to reduce the GI value of bread. A study conducted in 2020 showed that the GI value of regular white bread with 5% Cephalaria Syricia flour added decreased by 17%. Although there are in-vitro studies on the effects of Cephalaria Syricia in the literature, no clinical studies with published results have been found. From this point of view, this study is planned to investigate the effects of 0.2% Cephalaria Syricia flour added to bread (market name: İstanbul Halk Ekmek, Akdeniz Bread) on blood glucose and related hormones levels of individuals with diabetes and obesity and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Healthy group (n=20):

* 18-65 years of age, non-obese and non-diabetic healthy individuals
* OGTT is normal
* Body Mass Index (BMI)= 18.5-24.9 kg/m2

Diabetic group (n=20):

• Individuals aged between 18-65 years with Type 2 Diabetes

* Using only metformin
* BMI= 18.5-29.9 kg/m2

Obese group (n=20):

• 18-65 years of age, non-diabetic and obese individuals;

- BMI ≥ 30 kg/m2

Exclusion Criteria:

Individuals with

* Smoking
* Use Alcohol
* Pregnant
* Breastfeeding
* Those with chronic diseases (CKD, COPD, Malignancy,..)
* Using food supplements
* Using DPP-4 inhibitors and GLP-1release analog in the treatment of DM
* Professional athlete or excessive physical activity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Plasma GLP-1 levels changes | Through OGTT test completion, an average of 2 hours
  Change in baseline GLP-1 levels at 2 hours. Measured by plasma samples.
Plasma PYY levels changes | Through OGTT test completion, an average of 2 hours
  Change in baseline PYY levels at 2 hours. Measured by plasma samples.
Plasma Leptin levels changes | Through OGTT test completion, an average of 2 hours
  Change in baseline Leptin levels at 2 hours. Measured by plasma samples.
Plasma Ghrelin levels changes | Through OGTT test completion, an average of 2 hours
  Change in baseline Ghrelin levels at 2 hours. Measured by plasma samples.
Plasma IL-6 levels changes | Through OGTT test completion, an average of 2 hours
  Change in baseline IL-6 levels at 2 hours. Measured by plasma samples.
Plasma insulin levels changes | Through OGTT test completion, an average of 2 hours
  Change in baseline insulin levels at 2 hours. Measured by plasma samples.
Plasma glucose levels changes | Through OGTT test completion, an average of 2 hours
  Change in baseline glucose levels at 2 hours. Measured by plasma samples.
Plasma c-peptide levels changes | Through OGTT test completion, an average of 2 hours
  Change in baseline c-peptide levels at 2 hours. Measured by plasma samples.

SECONDARY OUTCOMES:
Plasma triglyceride levels changes | Through OGTT test completion, an average of 2 hours
  Change in baseline triglyceride levels at 2 hours. Measured by plasma samples.
Appetite regulation | Through OGTT test completion, an average of 2 hours
  Change in baseline appetite at 2 hours. Subjective appetite assessed with visual analog scales.
  The visual analog scale (VAS) is a psychometric response scale that can be used in questionnaires. It is a measurement tool for subjective characteristics or attitudes that cannot be measured directly.
  Visual analogue scales (VAS) were used to measure hunger (H), fullness (F), desire to eat (DtE), and prospective food consumption (PFC) scores (-s) immediately before consump- tion of test meal and at 60, 120, and 180 min later. The VAS-s were 100-mm straight line, and the patients were asked to make a vertical mark across this line corresponding to their concurrent feelings from 0 (not at all) to 100 (very) H, F, DtE, and PFC.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Faculty of Medicine, Department of Endocrinology and Metabolism, Istanbul, Capa, Turkey (Türkiye)